CLINICAL TRIAL: NCT01722370
Title: Can Muscle Dysfunction in COPD be Altered by Oxygenation in Patients With Intermittent Hypoxia on Exertion?
Brief Title: Ambulatory Oxygen Effects on Muscles in COPD
Acronym: OM-COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Heart of England NHS Trust (Other)
Responsible Party: Principal Investigator, Alice Turner, Dr, University of Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RG-11-132
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical air equivalent (Placebo Comparator): Oxygen-nitrogen mix equivalent to medical air when inhaled from a cylinder at 2l/min
  Interventions: Drug: Medical air equivalent
- Oxygen (Experimental): Ambulatory oxygen delivered at 2l/min on any activity performed by the patient, using a blinded cylinder
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen
  Arms: Oxygen
Drug: Medical air equivalent
  Arms: Medical air equivalent

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) may develop low oxygen levels, because of damage to their lungs. Long term oxygen therapy (LTOT) is given for at least 15 hours per day, and has established indications and benefits in COPD. However, the indications for and benefits from ambulatory oxygen supplementation (oxygen just when walking or exercising) are less well understood, in part due to heterogeneity of previous study designs, and lack of long term follow up. This is a pilot study of supplementary ambulatory oxygen in COPD, which allows us to ascertain mechanisms of disease by measuring their degree of systemic inflammation pre and post oxygen supplementation, and measuring changes in gene expression in muscles by means of microarray profiling. Secondly, our study will utilise follow up of clinical parameters including home activity monitoring to ascertain medium/long term benefits of oxygen supplementation in a real life setting. Our hypothesis is that exertional hypoxia results in muscle dysfunction and this could be prevented by oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD
* desaturation on exertion

Exclusion Criteria:

* using LTOT
* immobile for other reason than COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Gene expression pattern change between interventions in skeletal muscle biopsy | 12 weeks

SECONDARY OUTCOMES:
Six minute walk test distance | 12 weeks
Home activity level as measured by Actigraph | 6 and 12 weeks

OTHER OUTCOMES:
Blood gases | 12 weeks
Quality of life | 6 and 12 weeks
Anxiety and depression score | 12 weeks
Arterial stiffness | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice M Turner, Principal Investigator — University of Birmingham
Locations (1):
- Heart of England NHS Foundation Trust, Birmingham, West Midlands, United Kingdom